CLINICAL TRIAL: NCT00372190
Title: A Prospective and Comparative Study of the Performance of Tension Free Vaginal Mesh (Prolift) Versus Conventional Vaginal Prolapse Surgery in Recurrent Prolapse
Brief Title: Performance of Tension Free Vaginal Mesh (Prolift) Versus Conventional Vaginal Prolapse Surgery in Recurrent Prolapse.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Mariella Withagen, Principal Investigator, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P0609
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Results first posted 2017-07-03 (Actual); Last update posted 2017-07-03 (Actual); Status verified 2017-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; recurrence; mesh; complications; treatment
MeSH Terms: conditions — Pelvic Organ Prolapse; Recurrence | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesh surgery (Experimental): Trocar guided tension free vaginal mesh insertion by Prolift mesh kit
  Interventions: Device: Tensionfree vaginal mesh kit (Prolift)
- Conventional vaginal surgery (Active Comparator): Classical vaginal prolapse surgery (fascia plication)
  Interventions: Procedure: classic vaginal prolapse surgery (fascia plication)

INTERVENTIONS:
Device: Tensionfree vaginal mesh kit (Prolift) — Insertion of a tension free vaginal mesh using a Prolift mesh kit
  Other Names: Prolift mesh
  Arms: Mesh surgery
Procedure: classic vaginal prolapse surgery (fascia plication) — classic vaginal prolapse surgery (fascia plication) to correct Pelvic Organ prolapse
  Other Names: Conventional
  Arms: Conventional vaginal surgery

SUMMARY:
Pelvic organ prolapse is a common problem. A lot of women have surgery for prolapse. The recurrence rate op pelvic organ prolapse after surgical treatment is high. Placement of a mesh aims at reducing the recurrence rate, but mesh implants can cause complications.

This study is designed to determine the effectiveness of one type of mesh (tensionfree vaginal mesh; Prolift), compared with the standard prolapse surgery. A secondary objective is to track the complications of both procedures.

DETAILED DESCRIPTION:
Patients with recurrent prolapse after surgery can participate in this study. A total of 194 women will be included. At random 97 patients undergo a standard prolapse operation and 97 patients undergo an operation with the mesh. Evaluation will take place during surgery, at the postoperative visit after six weeks, and after six months and twelve months. Quality of life, degree of vaginal prolapse, subjective effectiveness, safety and incidence of complications will be evaluated.

An amendment to the original study has been approved by the Ethical Committee to examine long term outcome of this RCT at 7 years. This study was completed in december 2015.

ELIGIBILITY:
Inclusion Criteria:

* recurrent anterior and/or posterior prolapse POP-Q stage 2 or more
* patient has agreed to undergo implantation of TVM (prolift) or fascial plication
* patient is willing to return for follow-up evaluation at 6 weeks, 6 months and 12 months
* patient is willing to complete quality of life questionnaires at 6 and 12 months

Exclusion Criteria:

* patient is or wants to become pregnant
* patient has had previous synthetic mesh procedure (a previous mid-urethral sling procedure is NOT an exclusion criterion)
* patient has current urinary tract or vaginal infections
* patient has a blood coagulation disorder
* patient has a compromised immune system or any other condition that would compromise healing
* patient has renal insufficiency and/or upper urinary tract obstruction
* patient is unwilling or unable to return for evaluation
* patient has had previous irradiation
* patient has any malignancy
* patient has large ovarian cysts of large myoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2006-08; Primary Completion 2009-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariella ij Withagen, Drs., Principal Investigator — UMC St Radboud
Locations (13):
- Netherlands (13):
  - Gelre ziekenhuizen, Apeldoorn
  - Slysis Zorggroep, location Rijnstate, Arnhem
  - Reinier de Graaf Gasthuis, Delft
  - Medisch Spectrum Twente, Enschede
  - Groene Hart Ziekenhuis, Gouda
  - St. Antonius Ziekenhuis, Nieuwegein
  - UMC St Radboud, Nijmegen
  - Ikazia, Rotterdam
  - Refaja, Stadskanaal
  - St. Elisabeth hospital, Tilburg
  - Twee Steden Ziekenhuis, Tilburg
  - Zaans Medisch Centrum, Zaandam
  - Isala klinieken, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Withagen MI, Milani AL, den Boon J, Vervest HA, Vierhout ME. Trocar-guided mesh compared with conventional vaginal repair in recurrent prolapse: a randomized controlled trial. Obstet Gynecol. 2011 Feb;117(2 Pt 1):242-250. doi: 10.1097/AOG.0b013e318203e6a5. PMID 21252735
- [Derived] Milani AL, Damoiseaux A, IntHout J, Kluivers KB, Withagen MIJ. Long-term outcome of vaginal mesh or native tissue in recurrent prolapse: a randomized controlled trial. Int Urogynecol J. 2018 Jun;29(6):847-858. doi: 10.1007/s00192-017-3512-3. Epub 2017 Nov 22. PMID 29167974
- [Derived] Withagen MI, Milani AL, de Leeuw JW, Vierhout ME. Development of de novo prolapse in untreated vaginal compartments after prolapse repair with and without mesh: a secondary analysis of a randomised controlled trial. BJOG. 2012 Feb;119(3):354-60. doi: 10.1111/j.1471-0528.2011.03231.x. PMID 22239416

RESULTS

PARTICIPANT FLOW:
Groups:
- Mesh: Insertion of Tensionfree vaginal mesh (Prolift)
  Tensionfree vaginal mesh kit (Prolift): Insertion of a tension free vaginal mesh using a Prolift mesh kit.
  95 randomized for mesh, 2 refused surgery; 93 underwent mesh insertion
- Conventional: Classical vaginal prolapse surgery (fascia plication)
  classic vaginal prolapse surgery (fascia plication): classic vaginal prolapse surgery (fascia plication) to correct Pelvic Organ prolapse
  99 randomized to conventional surgery, 1 refused surgery for comorbidity, 1 died prior to surgery; 97 underwent conventional surgery
Period: Overall Study
Arm/Group | Mesh | Conventional
Started | 93 (95 were allocated to mesh group, however 2 never underwent any surgery) | 97 (99 were allocated to conventional arm, however 2 never underwent any surgery)
Completed | 90 | 96
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Mesh: Insertion of Tensionfree vaginal mesh (Prolift)
  Tensionfree vaginal mesh kit (Prolift): Insertion of a tension free vaginal mesh using a Prolift mesh kit
- Conventional: Classical vaginal prolapse surgery (fascia plication)
  classic vaginal prolapse surgery (fascia plication): classic vaginal prolapse surgery (fascia plication) to correct Pelvic Organ prolapse
- Total: Total of all reporting groups
Arm/Group | Mesh | Conventional | Total
Number analyzed (Participants) | 93 | 97 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] — age at randomization
  years | 64 (10.5) | 64 (10.2) | 64 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 97 | 190
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Prolapse by "Pelvic Organ Prolapse Quantification System" (POP-Q), at 12 Months
Description: Number of participants with anatomic failures defined as "Pelvic Organ Prolapse" (POP) stage II or higher
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Mesh | Conventional
Number analyzed (Participants) | 83 | 84
participants
  anatomic failures | 8 | 38
  anatomic success | 75 | 46
  no anatomic evaluation | 7 | 13
Statistical Analysis 1: Comparison: Mesh vs Conventional; Test type: Superiority or Other; p < 0.05, Chi-squared

2. Secondary Outcome: Mesh Exposure at 12 Months
Description: cumulative number of patients with mesh exposure at 12 months (if diagnosed at 6 weeks or 6 months and treated, the exposure is calculated at 12 months, even if the exposure was not there anymore)
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Mesh | Conventional
Number analyzed (Participants) | 93 | 97
participants | 14 | 0

3. Secondary Outcome: "Patient Global Impression of Improvement" (PGI-I) at 12 Months
Description: Number of participants with much to very much improvement compared to baseline
Time Frame: at 12 months
Measure: Number; unit: participants
Arm/Group | Mesh | Conventional
Number analyzed (Participants) | 84 | 88
participants | 54 | 54

4. Secondary Outcome: Bulge Symptoms
Description: Bulge symptoms defined as Prolapse domain score of the "Urogenital Distress Inventory" (UDI) at 12 months.
  Scores range from 0 (least/no bother) to 100 (maximum bother)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mesh | Conventional
Number analyzed (Participants) | 84 | 88
units on a scale | 6 (17) | 5 (17)

ADVERSE EVENTS:
Arm/Group | Mesh | Conventional
Serious Adverse Events (participants affected / at risk) | 8/93 | 2/97
Other Adverse Events (participants affected / at risk) | 25/93 | 11/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesh (N=93) | Conventional (N=97)
Bladder perforation (Renal and urinary disorders) | 2 (2) | 0 (0)
Repeat surgery for postoperative hematoma (Surgical and medical procedures) | 0 (0) | 1 (1)
Hematoma (Surgical and medical procedures) | 6 (6) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Mesh (N=93) | Conventional (N=97)
Mesh exposure (Surgical and medical procedures) | 14 (14) | 0 (0)
de novo dyspareunia (Reproductive system and breast disorders) | 3/37 (3) | 3/29 (3) — you can only develop de novo dyspareunia, if you had no dyspareunia before. therefore the number of women at risk is lower than in total
de novo SUI (Renal and urinary disorders) | 8/81 (8) | 8/88 (8) — you can only develop de novo SUI, if you had no SUI before, therefore the number is different from the total number of women at risk

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes